CLINICAL TRIAL: NCT03448640
Title: Efficiency and Safety of Phenylephrine and Tropicamide Used in Premature Retinopathy
Brief Title: Efficacy of Mydriatic Drops in Premature Infants
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Atilla Alpay, Asociate Pofessor Atilla Alpay, Bulent Ecevit University
Other Study IDs: BulentEU
Record Dates: First submitted 2018-02-15; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Tropicamide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Drug used in the examination of premature infants. — to investigate side effects of eye drops used
  Other Names: Tropicamide and mydfline used

SUMMARY:
Because of the neonatologists reported that some infants had suffered from vomiting, bradycardia, hypotonia, and aspiration risk about 30-60 minutes after the fundus examination in the intensive care unit. The investigators observed the pupil dilation effects and side effects of tipple instillation of phenylephrine 2.5% plus tropicamide 0.5% ophthalmic drop combination which the investigators routinely used in ROP examination.

DETAILED DESCRIPTION:
Purpose: To determine effect and vital change after topical application of phenylephrine 2.5% and tropicamide 0.5% three times for retinopathy of prematurity (ROP) examination in preterm infants.

Methods: Pupillary diameter, blood pressure, pulse rate, and oxygen saturation were monitored before, and after up to 24 hours 60 ROP screening examinations.

ELIGIBILITY:
Inclusion Criteria:

* Infants who were first ROP examinations
* infants born before 32 weeks.

Exclusion Criteria:

* Developmental ocular and/or systemic anomalies.
* Drug use that can affect vital values
* Unstable general condition
* Food intolerance
* Recurrent vomiting.

Ages: 32 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — neonatal
Study Population: tertiary health center in the west Black Sea region
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
The mean pupillary diameter | an average of 1 year
  will be measured with a ruler after 60 minutes instillation of mydriatic

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spencer R. Long-term visual outcomes in extremely low-birth-weight children (an American Ophthalmological Society thesis). Trans Am Ophthalmol Soc. 2006;104:493-516. PMID 17471358
- [Background] Sindel BD, Baker MD, Maisels MJ, Weinstein J. A comparison of the pupillary and cardiovascular effects of various mydriatic agents in preterm infants. J Pediatr Ophthalmol Strabismus. 1986 Nov-Dec;23(6):273-6. doi: 10.3928/0191-3913-19861101-04. PMID 3454368
- [Background] Clarke WN, Hodges E, Noel LP, Roberts D, Coneys M. The oculocardiac reflex during ophthalmoscopy in premature infants. Am J Ophthalmol. 1985 Jun 15;99(6):649-51. doi: 10.1016/s0002-9394(14)76029-5. PMID 4014388
- [Background] Lim DL, Batilando M, Rajadurai VS. Transient paralytic ileus following the use of cyclopentolate-phenylephrine eye drops during screening for retinopathy of prematurity. J Paediatr Child Health. 2003 May-Jun;39(4):318-20. doi: 10.1046/j.1440-1754.2003.00144.x. PMID 12755944
- [Background] Bonthala S, Sparks JW, Musgrove KH, Berseth CL. Mydriatics slow gastric emptying in preterm infants. J Pediatr. 2000 Sep;137(3):327-30. doi: 10.1067/mpd.2000.107842. PMID 10969255
- [Background] Chien DS, Homsy JJ, Gluchowski C, Tang-Liu DD. Corneal and conjunctival/scleral penetration of p-aminoclonidine, AGN 190342, and clonidine in rabbit eyes. Curr Eye Res. 1990 Nov;9(11):1051-9. doi: 10.3109/02713689008997579. PMID 1982760
- [Background] Thanathanee O, Ratanapakorn T, Morley MG, Yospaiboon Y. Lower conjunctival fornix packing for mydriasis in premature infants: a randomized trial. Clin Ophthalmol. 2012;6:253-6. doi: 10.2147/OPTH.S28714. Epub 2012 Feb 15. PMID 22368443
- [Background] Cohen AM, Cook N, Harris MC, Ying GS, Binenbaum G. The pain response to mydriatic eyedrops in preterm infants. J Perinatol. 2013 Jun;33(6):462-5. doi: 10.1038/jp.2012.149. Epub 2012 Dec 13. PMID 23238569
- [Background] Ballabh P. Intraventricular hemorrhage in premature infants: mechanism of disease. Pediatr Res. 2010 Jan;67(1):1-8. doi: 10.1203/PDR.0b013e3181c1b176. PMID 19816235
- [Background] Wilkinson AR, Haines L, Head K, Fielder AR. UK retinopathy of prematurity guideline. Early Hum Dev. 2008 Feb;84(2):71-4. doi: 10.1016/j.earlhumdev.2007.12.004. No abstract available. PMID 18280404
- [Result] Laws DE, Morton C, Weindling M, Clark D. Systemic effects of screening for retinopathy of prematurity. Br J Ophthalmol. 1996 May;80(5):425-8. doi: 10.1136/bjo.80.5.425. PMID 8695564
- [Result] Lees BJ, Cabal LA. Increased blood pressure following pupillary dilation with 2.5% phenylephrine hydrochloride in preterm infants. Pediatrics. 1981 Aug;68(2):231-4. PMID 7267230
- [Result] Isenberg S, Everett S, Parelhoff E. A comparison of mydriatic eyedrops in low-weight infants. Ophthalmology. 1984 Mar;91(3):278-9. doi: 10.1016/s0161-6420(84)34303-2. PMID 6546977
- [Result] Alpay A, Ermis B, Ugurbas SC, Battal F, Sagdik HM. The local vasoconstriction of infant's skin following instillation of mydriatic eye drops. Eur J Clin Pharmacol. 2010 Nov;66(11):1161-4. doi: 10.1007/s00228-010-0890-6. Epub 2010 Sep 11. PMID 20835704
- [Result] Khoo BK, Koh A, Cheong P, Ho NK. Combination cyclopentolate and phenylephrine for mydriasis in premature infants with heavily pigmented irides. J Pediatr Ophthalmol Strabismus. 2000 Jan-Feb;37(1):15-20. doi: 10.3928/0191-3913-20000101-05. PMID 10714690
- [Result] Lux AL, Degoumois A, Barjol A, Mouriaux F, Denion E. Combination of 5% phenylephrine and 0.5% tropicamide eyedrops for pupil dilation in neonates is twice as effective as 0.5% tropicamide eyedrops alone. Acta Ophthalmol. 2017 Mar;95(2):165-169. doi: 10.1111/aos.13175. Epub 2016 Aug 13. PMID 27519933
- [Result] Ogut MS, Bozkurt N, Ozek E, Birgen H, Kazokoglu H, Ogut M. Effects and side effects of mydriatic eyedrops in neonates. Eur J Ophthalmol. 1996 Apr-Jun;6(2):192-6. doi: 10.1177/112067219600600218. PMID 8823596
- [Result] Mitchell AJ, Green A, Jeffs DA, Roberson PK. Physiologic effects of retinopathy of prematurity screening examinations. Adv Neonatal Care. 2011 Aug;11(4):291-7. doi: 10.1097/ANC.0b013e318225a332. PMID 22123352
- [Result] Patel AJ, Simon JW, Hodgetts DJ. Cycloplegic and mydriatic agents for routine ophthalmologic examination: a survey of pediatric ophthalmologists. J AAPOS. 2004 Jun;8(3):274-7. doi: 10.1016/j.jaapos.2004.01.004. PMID 15226730
- [Result] Rush R, Rush S, Nicolau J, Chapman K, Naqvi M. Systemic manifestations in response to mydriasis and physical examination during screening for retinopathy of prematurity. Retina. 2004 Apr;24(2):242-5. doi: 10.1097/00006982-200404000-00009. PMID 15097885
- [Result] Neffendorf JE, Mota PM, Xue K, Hildebrand GD. Efficacy and safety of phenylephrine 2.5% with cyclopentolate 0.5% for retinopathy of prematurity screening in 1246 eye examinations. Eur J Ophthalmol. 2015 May-Jun;25(3):249-53. doi: 10.5301/ejo.5000540. Epub 2014 Nov 14. PMID 25449644
- [Result] Mitchell A, Hall RW, Erickson SW, Yates C, Lowery S, Hendrickson H. Systemic Absorption of Cyclopentolate and Adverse Events After Retinopathy of Prematurity Exams. Curr Eye Res. 2016 Dec;41(12):1601-1607. doi: 10.3109/02713683.2015.1136419. Epub 2016 May 9. PMID 27159349
- [Result] Anand KJ. Clinical importance of pain and stress in preterm neonates. Biol Neonate. 1998;73(1):1-9. doi: 10.1159/000013953. PMID 9458936
- [Result] Belda S, Pallas CR, De la Cruz J, Tejada P. Screening for retinopathy of prematurity: is it painful? Biol Neonate. 2004;86(3):195-200. doi: 10.1159/000079542. Epub 2004 Jul 5. PMID 15240989
- [Derived] Alpay A, Canturk Ugurbas S, Aydemir C. Efficiency and safety of phenylephrine and tropicamide used in premature retinopathy: a prospective observational study. BMC Pediatr. 2019 Nov 6;19(1):415. doi: 10.1186/s12887-019-1757-3. PMID 31690284